CLINICAL TRIAL: NCT06326242
Title: Toward a Patient-centered Early Drug Development in Oncology: What Unmet Need for the Patients? A Focus on the Social Determinants of Health in Phase 1 Clinical Trials
Brief Title: What Unmet Need for the Patients?A Focus on the Social Determinants of Health in Phase 1 Clinical Trials
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1648
Record Dates: First submitted 2024-03-13; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor
MeSH Terms: interventions — PMEPA1 protein, human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Solid Tumor: Phase 1 patient with solid tumor
  Interventions: Other: Solid Tumor

INTERVENTIONS:
Other: Solid Tumor — The study focuses on defining the problem of geographical accessibility of patients to the Phase 1 facility of the European Institute of Oncology, based on anonymized data extraction from the enrolled patient database, to evaluate national territorial disparities in access to innovative experimental therapies, in relation to various socioeconomic determinants. Finally, relevant information on psychological factors for participation in clinical trials will also be collected.

SUMMARY:
An observational prospective study of patients enrolled and treated with experimental drugs in Phase I studies.

DETAILED DESCRIPTION:
The study focuses on defining the problem of geographical accessibility of patients to the Phase 1 facility of the European Institute of Oncology, based on an anonymized extraction of data from the enrolled patient database, to assess national territorial disparities in access to innovative experimental therapies, in relation to various socioeconomic determinants. Finally, information on relevant psychological factors for participation in clinical trials will also be collected.

ELIGIBILITY:
Inclusion Criteria :

* Patient with a histological or cytological diagnosis of solid or hematological tumor.
* Age ≥ 18 years.
* Patient enrolled in a phase 1 and early phase 2 study at our institution.
* The patient has received at least 1 administration of the experimental drug under study in the early phase trial.

Exclusion Criteria :

- Patients treated in phase 1 trials at other institutions, even if referred to our division or receiving standard therapies at IEO but outside of clinical trials, are not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient enrolled in a phase 1 and early phase 2 study at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The geographical accessibility of patients attending the Phase 1 facility of the European Institute of Oncology (IEO). | 1 year
  The primary endpoint is estimating the geographical distance from the enrolled patients' residences to the European Institute of Oncology (IEO), evaluating patients from the Lombardy region versus those from other regions with an assessment by geographical cluster: north, central, south, and islands, in order to define any preferential trajectories or recurring patterns.

SECONDARY OUTCOMES:
The characterization of enrolled patients involves assessing their participation in clinical trials | 1 year
  The enrolled patients will be characterized based on psychological factors included in the study. These factors include: patient attitudes, perceived social norms, and perceived control over participation in clinical studies; doctor-patient relationship; study awareness; evaluation of their own decision to participate in the study
The characterization of enrolled patients based on therapeutic compliance. | 1 year
  The evaluation of compliance with protocol procedures unrelated to the administration of the experimental drug, such as pharmacokinetic sampling and study biopsies
The protocol prescriptions in relation to socioeconomic and geographical determinants. | 1 year
  The correlations with metrics of geographic accessibility and income per area of origin will be explored in accordance with ISTAT (Italian National Statistics Institute) data, where applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Profeta, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of oncology, Milan, Italy